CLINICAL TRIAL: NCT01073787
Title: Single-blind, Placebo-challenge Study of Intravenous Fluid Hydration in the Management of Pediatric Migraine in the Emergency Department
Brief Title: Intravenous Fluid for Pediatric Migraine in the Emergency Department
Acronym: EDMigraine3
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00008034
Record Dates: First submitted 2010-02-22; First posted 2010-02-23 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Migraine; Headache
Keywords: migraine; headache; pediatric; children; Emergency Department
MeSH Terms: conditions — Migraine Disorders; Headache; Emergencies | interventions — Saline Solution; Sodium Chloride; Water

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal saline (Active Comparator)
  Interventions: Drug: Normal saline
- Normal saline and possible medication (Experimental)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Normal saline — 10 ml/kg of normal saline will be administered over 30 minutes
  Other Names: 0.9% sodium chloride and water

SUMMARY:
The purpose of this study is to evaluate the effect of intravenous fluid (0.9% sodium chloride and water) alone on headache pain in children with migraine visiting the Emergency Department.

DETAILED DESCRIPTION:
Migraine is a common and disabling disorder for children. The pain may be severe and relatively few effective medications are approved for use in children. The Emergency Department (ED) remains an important resource for children suffering from migraine whom have not responded to their usual therapy. While a number of effective intravenous therapies have been studied in adults, there has been only one such study in children. As such, emergency physicians have little or no information about the safety and efficacy of these medications in children. However, the conduct of clinical trials where pain is the outcome measure is often limited by a high placebo-response rate. The expectation of treatment can significantly alter the response to medications especially when pain severity is the outcome measure. Moreover, the investigators have found that intravenous fluid alone may help to treat migraine headache in children. The investigators propose a study to examine the response to intravenous fluid hydration as initial therapy comparing a group with expectation of medication and another group without the initial expectation of medication. The results of the study will help to estimate the rate of response to intravenous fluid and to evaluate the placebo-effect (i.e. expectation of treatment) in studies of migraine treatment in the ED. Exposure to additional and possibly unnecessary medications will thus be minimized and the results of future trials more definitive on the effect of the study medication.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of migraine or probable migraine (with or without aura) per the International Classification of Headache Disorders (2nd edition)
* Visiting the Emergency Department for migraine treatment
* Emergency Department physician has chosen to administer intravenous medication
* Has taken usual therapy at home or at least one does of either ibuprofen or acetaminophen in the Emergency Department

Exclusion Criteria:

* Other probable cause for headache (e.g. ventriculoperitoneal shunt, neoplasm, intracranial cyst)
* Head trauma causing loss of consciousness within 1 week of presentation
* Fever (temperature > 38.5 oC)
* Signs or symptoms of meningitis

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Headache pain | 30 minutes
  Pain will be assessed using three measures: (1) Nine Faces Pain scale; (2) Visual Analogue Scale; and (3) Four categories (none, mild, moderate, or severe)

SECONDARY OUTCOMES:
Nausea | 30 minutes
  Severity will be assessed using: (1) Visual Analogue Scale; (2) Four categories (none, mild, moderate, severe)
Vomiting | 30 minutes
Use of rescue medication | 24 hours
  Use of any rescue medication after leaving the Emergency Department
Headache recurrence | 24 hours
  Recurrence or worsening of headache after leaving the Emergency Department
Return to Emergency Department | 24 hours
  Return to Emergency Department for treatment of migraine within 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence P Richer, MD, MSc, Principal Investigator — University of Alberta
Locations (1):
- Stollery Children's Hospital Emergency Department, Edmonton, Alberta, Canada

REFERENCES:
- [Result] Richer L, Craig W, Rowe B. Randomized controlled trial of treatment expectation and intravenous fluid in pediatric migraine. Headache. 2014 Oct;54(9):1496-505. doi: 10.1111/head.12443. Epub 2014 Aug 28. PMID 25168404